CLINICAL TRIAL: NCT03158922
Title: The BARCODE 1 Pilot Study: The Use of Genetic Profiling to Guide Prostate Cancer Targeted Screening
Brief Title: The BARCODE 1 Pilot Study
Acronym: BARCODE1Pilot
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4130
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1: Caucasian men aged 55-69 to undergo genetic profiling.
  Interventions: Genetic: Genetic SNP profiling
- Stage 2: Men from Stage 1 identified as having a higher genetic risk score (top 10%) for prostate cancer.
  Interventions: Genetic: Genetic SNP profiling; Other: Prostate cancer screening; Procedure: Prostate biopsy

INTERVENTIONS:
Genetic: Genetic SNP profiling — Genetic SNP profiling of known prostate cancer predisposition SNPs will be performed on DNA extracted from saliva samples.
Other: Prostate cancer screening — Prostate cancer screening in the form of PSA testing will be offered to all men who have a benign biopsy result for five years in order to track development of cancer in the future.
  Groups: Stage 2
Procedure: Prostate biopsy — Prostate biopsy will be offered to men identified within the top 10% genetic risk score profile.
  Other Names: TRUS Biopsy
  Groups: Stage 2

SUMMARY:
BARCODE 1 is a screening study designed to investigate the role of genetic profiling for targeting population prostate cancer screening. This study forms a pilot of 300 men, with the view to continue to a future study of 5000 men.

DETAILED DESCRIPTION:
The BARCODE 1 study aims to evaluate genetic profiling using the known 170 prostate cancer (PrCa) risk single-nucleotide polymorphisms (SNPs) as a means of offering targeted screening for PrCa in men at a genetically higher risk. Initially, 300 men will be recruited via participating General Practices (GPs). Men aged 55-69 years who are likely to be eligible for the study will be identified by GPs from medical records. Participants will be contacted via invitation letters from GPs and if interested in the study will be asked to fill in a questionnaire to confirm eligibility to participate. This questionnaire can be completed in hard copy and men will also be given the option to fill in an online version. If eligible, men will then be sent a DNA collection saliva kit. DNA from saliva will be analysed with SNP profiling for the known 170 clinically relevant SNPs. Men with a genetic risk equivalent to the top 10% of the population distribution (approximately 30 men in total) will be invited for a transrectal ultrasound (TRUS) prostate biopsy, plus further biological samples. Biopsy results will be correlated with the genetic score. Prostate-specific antigen (PSA) and other biomarkers will be integrated into results to assess combined effects of genetic score and markers.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 55-69 years
* Caucasian ethnicity
* World Health Organisation (WHO) performance status 0-2
* Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule

Exclusion Criteria:

* Non-Caucasian ethnicity (including mixed race or Jewish)
* Previous diagnosis of cancer with a life-expectancy of less than five years
* Prostate biopsy in the past year
* Previous diagnosis of prostate cancer
* Co-morbidities making prostate biopsy risk unacceptable (anticoagulants or antiplatelet medication like Warfarin or Clopidogrel, poorly controlled diabetes or cardiovascular disease)

Ages: 55 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men of Caucasian ethnicity (not Mixed race or Jewish), aged 55 - 69 years, willing to undergo genetic SNP profiling.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of SNP genetic risk score with prostate biopsy results. | 5 years

SECONDARY OUTCOMES:
Incidence and aggressiveness of PrCa in men within the top 10% of the genetic score. | 5 years
Association of the biomarker profile with genetic score and biopsy results. | 5 years
Use of genetic profiling to target prostate cancer screening in a clinical environment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, FRCP, FRFR, Principal Investigator — Institute of Cancer Research and Royal Marsden Hospital
Locations (1):
- Institute of Cancer Research and Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Data Access Committee.